CLINICAL TRIAL: NCT05204797
Title: Efficacy of Robot-assisted Technique vs Conventional Technique in Preventing Early Micromobilisation After Unicompartmental Knee Arthroplasty: a Controlled Randomized Trial
Brief Title: Efficacy of Robot-assisted Technique vs Conventional Technique in Preventing Early Micromobilisation After UKA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Principal Investigator, Stefano Zaffagnini, Head of Orthopaedics and Traumatology II Clinic, Istituto Ortopedico Rizzoli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: RSA UNI CORI
Record Dates: First submitted 2021-09-27; First posted 2022-01-24 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Loosening, Prosthesis
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: Two blinded groups operated via robotic-assisted surgery (1st arm) or conventional technique (2nd arm).
Who Masked: Participant
Masking Description: At the research office of health professions at IRCCS Istituto Ortopedico Rizzoli in Bologna, Italy (coordinating centre), a block of 5 randomisation list using the site "www.randomisation.com" will be generated. A sequence of opaque envelopes will be set up with a sequential number on the outside. A label will be placed iside the envelope that will contain the words "CORI" or "STANDARD", according to the sequence indicated by the generated list. Envelopes will be always sealed at the Research Centre and the list kept under lock. The envelopes will be placed in a dedicated box and delivered to the studio manager.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Robot-assisted UKA (Experimental): Unicompartmental knee replacement (Journey II UKA, Smith and Nephew, USA) positioned via CORI surgical system (Smith & Nephew, USA).
  Interventions: Procedure: Robot-assisted UKA
- Standard technique UKA (Active Comparator): Unicompartmental knee replacement (Journey II UKA, Smith and Nephew, USA) positioned via standard technique.
  Interventions: Procedure: Standard technique UKA

INTERVENTIONS:
Procedure: Robot-assisted UKA — Cemented unicompartmental knee arthroplasty via mini-invasive medial approach and robotic assistance. Tourniquet will be used in all patients.
  Other Names: CORI Surgical System, Smith and Nephew
  Arms: Robot-assisted UKA
Procedure: Standard technique UKA — Cemented unicompartmental knee arthroplasty via mini-invasive medial approach and standard technique. Tourniquet will be used in all patients.
  Arms: Standard technique UKA

SUMMARY:
The purpose of this study is to compare the percentage of early micromibilisation in unicompartmental knee arthroplasties in robot-assisted technique vs standard technique.

DETAILED DESCRIPTION:
The purpose of the study is to compare the percentage of early micromobilisation by static radiostereometric analysis (RSA) - primary outcome, gait analysis by inertial sensors to assess gait kinematics, and clinical perdormance measured by american knee society score (AKSS), oxford knee score (OKS), patient satisfaction score (PSS) and EQ5-D - secondary outcomes, among 2 groups of patients, of 25 individuals each, whi undergo medial unicompartmental knee arthroplasty.

The first group will be operated with a robot-assisted technique (with CORI Surgical System, Smith and Nephew, USA), the other with standard technique and the same implant (Journey UNI II, Smith and Nephew, USA).

The study will be a randomized and controlled blind superiority trial. Patients will not be informed about performing the surgery with one technique or the other in order to avoid potential biases in the data analysis.

Patients will be recruited at the orthoaedic and traumatologic 2nd clinica (head prof S. Zaffagnini) at IRCSS Istituto Ortopedico Rizzoli in Bologna, Italy.

ELIGIBILITY:
Inclusion Criteria:

* Unicompartmental Knee Arthrosis
* Femoral condyles or medial tibial plate osteonecrosis
* Healthy anterior cruciate ligament, posterior cruciate ligament and collateral ligaments of the affected knee
* Post traumatic loss of joint configuration
* Moderate varism deformity
* Patients between 50 and 80 years old
* Patients able to undergo a 2-year follow up after surgery

Exclusion Criteria:

* Bi or Tricompartmental arthrosis
* Unhealty anterior or posterior cruciate ligaments or collateral ligaments
* Patients with neuromuscolar, degenerative and joint-related conditions
* Patients younger than 50
* Patients older than 80
* Patients unable to undergo a 2-year follow up after surgery

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Static radiostereometric analysis (RSA) | Within 7 days from surgery, during hospitalisation
  Dual X-Ray simultaneous evaluation of micromobilisation via radiopaque markers and software comparison
Static radiostereometric analysis (RSA) | 3 months
  Dual X-Ray simultaneous evaluation of micromobilisation via radiopaque markers and software comparison
Static radiostereometric analysis (RSA) | 6 months
  Dual X-Ray simultaneous evaluation of micromobilisation via radiopaque markers and software comparison
Static radiostereometric analysis (RSA) | 12 months
  Dual X-Ray simultaneous evaluation of micromobilisation via radiopaque markers and software comparison
Static radiostereometric analysis (RSA) | 24 months
  Dual X-Ray simultaneous evaluation of micromobilisation via radiopaque markers and software comparison

SECONDARY OUTCOMES:
Gait analysis via inertial sensors | Within 7 days from surgery, during hospitalisation
  Inertial sensors (Awinda, Xsens Technologies and Gwalk, BTS engineering) will be placed on the patients then performed walking under VICON cameras analysis.
Gait analysis via inertial sensors | 6 months
  Inertial sensors (Awinda, Xsens Technologies and Gwalk, BTS engineering) will be placed on the patients then performed walking under VICON cameras analysis.
Gait analysis via inertial sensors | 24 months
  Inertial sensors (Awinda, Xsens Technologies and Gwalk, BTS engineering) will be placed on the patients then performed walking under VICON cameras analysis.
American Knee Society score | Pre-operatively, then at 3, 6, 12 and 24 months follow-up
  Used to test knee function by the investigator: it has a clinical and a functional part
Oxford Knee Score | Pre-operatively, then at 3, 6, 12 and 24 months follow-up
  Consists of 12 questions to be filled by the patient to assess how the prosthesis affect activities of daily living.
Patient Satisfaction Score | Pre-operatively, then at 3, 6, 12 and 24 months follow-up
  A short personal questionnaire that assesses subjective satisfaction after surgery
EQ5-D questionnaire | Pre-operatively, then at 3, 6, 12 and 24 months follow-up
  a questionnaire filled by the patient assessing the overall health of the subject. It is a test used to assess quality of life index.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Zaffagnini, Prof., Principal Investigator — IRCCS Istituto Ortopedico Rizzoli; Giulio Maria Marcheggiani Muccioli, Prof., Study Director — IRCCS Istituto Ortopedico Rizzoli; Stefano Fratini, Dr., Study Chair — IRCCS Istituto Ortopedico Rizzoli; Stefano Di Paolo, Eng., Study Chair — University of Bologna; Laura Bragonzoni, Dr., Study Chair — University of Bologna; Raffaele Zinno, Dr., Study Chair — University of Bologna; Giuseppe Barone, Dr., Study Chair — University of Bologna
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No
No sharing planned